CLINICAL TRIAL: NCT06307132
Title: A Study on the Correlation of Drug Metabolism, Excretion, and Human Body Composition Based on the Bioequivalence Trial of Aximus Capsules
Brief Title: Drug Metabolism, Excretion, and Human Body Composition of Aximus Capsules
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, TING LI, chief physician, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2024-03-106
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Bioequivalence Trial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test preparation
  Interventions: Other: Aximus capsules（test）
- reference preparation
  Interventions: Drug: Aximus capsules（reference）

INTERVENTIONS:
Other: Aximus capsules（test） — Aximus capsules test preparation
  Groups: test preparation
Drug: Aximus capsules（reference） — Aximus capsules reference preparation
  Groups: reference preparation

SUMMARY:
This project will be based on the bioequivalence test of Aximus capsules, measuring the body composition indicators of healthy subjects before and after medication, and collecting urine samples from subjects at different time periods after medication, measuring urine drug concentration, calculating urine excretion, analyzing the individualized differences in metabolism and excretion of Aximus capsules under different health states of human components, and providing guidance for clinical precision medication.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and non-pregnant non-lactating women who successfully participated in the bioequivalence test of acylimus capsules；
2. Signed the informed consent form, and fully understood the content, process and risks of this research, and be able to communicate well with the researchers.

Exclusion Criteria:

1. Female subjects who are menstruating (which may affect urine sample collection);
2. The subjects may not be able to complete this study for other reasons or may not be suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Excretion volume | Within 12 hours after taking medication
  drug concentration in urine

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of WMU Phase l Clinical Trial Unit /Center Of Bioequivalence Study, Wenzhou, China

IPD SHARING:
Plan to Share IPD: Undecided